CLINICAL TRIAL: NCT07268885
Title: The Efficacy and Safety of Platelet Rich Plasma Spinoplasty in the Management of Lower Back Pain Due to Multiple Pathologies: A Quasi-Experimental Study
Brief Title: PRP Spinoplasty for Chronic Low Back Pain With Multiple Pathologies: A Quasi-Experimental Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allmed Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Mustafa A Hammad, Medical Director and Principal Investigator, Allmed Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC.MRC.March4222024
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Lower Back Pain Chronic; Lumbar Disc Disease; Facet Joint Arthritis
Keywords: Platelet Rich Plasma; Lower back pain; lumbar disc disease
MeSH Terms: conditions — Intervertebral disc disease; Low Back Pain | interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with chronic low back pain secondary to lumbar disc disease and facet arthropathy (Experimental): The study population consisted of 35 adult patients with a diagnosis of chronic low back pain secondary to lumbar disc disease and facet arthropathy, with an associated component of muscular spasm. Diagnoses were confirmed by an interventional pain specialist based on a detailed medical history, physical examination, and magnetic resonance imaging (MRI) findings.
  Interventions: Biological: Spinoplasty with Platelet Rich Plasma

INTERVENTIONS:
Biological: Spinoplasty with Platelet Rich Plasma — The patient received a procedure called "Spinoplasty" which interlaminar epidural, facet joints and trigger point injection with Platelet Rich Plasma (PRP).
  Other Names: Epidural injection; Facet Joint Injection; Trigger Point Injection

SUMMARY:
This study aimed to evaluate the efficacy and safety of a comprehensive, multi-target injection protocol, termed 'PRP Spinoplasty,' for managing chronic LBP stemming from concurrent lumbar disc and facet joint disease with associated muscle spasms.

DETAILED DESCRIPTION:
A quasi-experimental study was conducted on 29 patients with chronic LBP who failed conservative therapy. The PRP Spinoplasty protocol involved a single-session, fluoroscopy-guided administration of autologous PRP to the interlaminar epidural space, affected facet joints, and paraspinal muscle trigger points. Outcomes were assessed using the Numeric Pain Scale (NPS), Oswestry Disability Index (ODI), and Single Assessment Numeric Evaluation (SANE) at baseline and at 1 week, 1 month, 3 months, and 6 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes; ages between 18 and 80 years.
* Lower back pain consistent with lumbosacral radiculopathy, facet arthropathy, and muscle spasms.
* MRI-confirmed lumbar spine pathology (disc disease and/or facet arthropathy).
* Failure to respond to at least 3 months of conservative therapy (NSAIDS and physical therapy).
* Pain score ≥ 6; on the 10-point Numeric Pain Scale (NPS) at baseline.

Exclusion Criteria:

* Presence of local or systemic infection, or fever.
* Diagnosed with cancer within the past 12 months.
* Unable to give a consent.
* History of spinal deformity such as fracture, or severe spinal stenosis causing neurological deficit.
* Presence of lower extremity weakness or urinary tract symptoms related to spinal pathology.
* Previous spinal decompression or fusion surgery at the treatment level.
* Receipt of any spine injection within the previous 12 months.
* Use of NSAIDs within 2 weeks prior to, or 6 weeks following the procedure.
* Use of corticosteroids within 6 weeks prior, or after the procedure.
* Use of anticoagulation or antiplatelet drugs (excluding low-dose Aspirin).
* History of blood disorders.
* History of any major surgery within the past 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Quantifying pain intensity using Numeric Pain Scale (NPS) | 0-6 months
  An 11-point scale (0 = no pain, 10 = worst imaginable pain) used to quantify pain intensity
Assessing level of functional disability using Oswestry Disability Index (ODI) | 0-6 months
  A 10-item questionnaire assessing the level of functional disability due to low back pain. Scores are calculated from a raw point score of 0-52, with lower scores indicating less disability. The raw score corresponds to the following disability levels: 0-4 points (No disability), 5-14 points (Mild disability), 15-24 points (Moderate disability), 25-34 points (Severe disability), and 35-52 points (Completely disabled)
Assessing patient's condition using Single Assessment Numeric Evaluation (SANE) | 0-6 months
  A patient-reported global assessment score where patients rate their condition on a scale of 0-100%, comparing their current status to their pre-injury baseline

SECONDARY OUTCOMES:
Assessing adverse events from treatment | 0-6 months
  Adverse events were monitored and systematically recorded at each follow-up contact. Patients were asked about any potential complications, including but not limited to severe post-procedural pain, signs of infection (fever, erythema, swelling), new or worsening neurological symptoms, or any other unexpected medical events. we use a checklist of possible complications questionnaire that patients were asked about during follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa A Hammad, MD, Principal Investigator — Allmed Medical Center
Locations (1):
- Allmed Medical Center, Ramallah, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the reported results (de-identified clinical and demographic variables) will be made available to qualified researchers upon reasonable request. All shared data will be fully anonymized in accordance with institutional and ethical guidelines. No direct identifiers will be included.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available following the publication of the primary manuscript. The data will remain available for a period of 5 years following publication.
Access Criteria: Data will be shared with qualified academic researchers for legitimate research purposes (e.g., meta-analysis, verification of findings). Requests must be sent to the corresponding author (Mustafa A. Hammad at neuro711@gmail.com). Requesters will need to provide a brief research proposal and sign a data use agreement (DUA) to ensure patient confidentiality is maintained.

REFERENCES:
- See also: Machado ES, Ambach MA, Caldas JM, Wei JJ, Bredemeier M. Personalized multitarget biologic injection in the spine: prospective case series of multitarget platelet-rich plasma for low back pain. Regen Med. 2022;17(1):11-22 — https://pubmed.ncbi.nlm.nih.gov/34907784/
- See also: Zhang X et al. The Clinical Efficacy of Platelet-Rich Plasma Injection Therapy versus Different Control Groups for Chronic Low Back Pain: A Network Meta-Analysis of Randomized Controlled Trials. J Pain Res. 2024;17:1077-1089 — http://doi.org/10.2147/JPR.S444189
- See also: Muthu S, Viswanathan VK, Gangadaran P. Is platelet-rich plasma better than steroids as epidural drug of choice in lumbar disc disease with radiculopathy? Meta-analysis of randomized controlled trials. Exp Biol Med. 2025;Volume 250 — http://doi.org/10.3389/ebm.2025.10390
- See also: Mohammed S, Yu J. Platelet-rich plasma injections: an emerging therapy for chronic discogenic low back pain. J Spine Surg. 2018;4(1):115 — http://doi.org/10.21037/jss.2018.03.04
- See also: Baltzer AW, Enneper J, Baltzer LM, Godde G. Platelet Rich Plasma for the Therapy of the Lumbar Facet Joint Syndrome: A Prospective Study About CT-Guided Facet Joint Injections With PRP Compared to Local Anesthetics. Orthop Rev (Pavia). 2025;17:141416 — http://pubmed.ncbi.nlm.nih.gov/40823278/
- See also: Xuan Z, Yu W, Dou Y, Wang T. Efficacy of Platelet-rich Plasma for Low Back Pain: A Systematic Review and Meta-analysis. J Neurol Surgery, Part A Cent Eur Neurosurg. 2020;81(6):529-534 — http://doi.org/10.1055/S-0040-1709170